CLINICAL TRIAL: NCT06495632
Title: Scheduled or As Needed Regimen? a Pilot Feasibility Study on Multimodal Pain Control and Post-Operative Pain
Brief Title: Scheduled or As Needed Pain Regimen?
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Cape Fear Valley Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1185-24
Record Dates: First submitted 2024-07-02; First posted 2024-07-11 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Pain, Postoperative
Keywords: surgery; acute pain; post-operative pain
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Ibuprofen; Narcotics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- scheduled pain regimen (Active Comparator): This group will receive post-operative pain medications including narcotics for 2-3 days (Oxycodone/Acetaminophen 5mg/325mg, Hydrocodone/Acetaminophen 5mg/325mg, Hydromorphone 2mg, or Tramadol 50mg) every 4 hours and 800 mg Motrin for 10 days every 8 hours on a fixed time/day schedule.
  Interventions: Drug: Motrin and narcotic
- as needed pain regimen (Experimental): This group will receive post-operative pain medications including narcotics for 2-3 days (Oxycodone/Acetaminophen 5mg/325mg, Hydrocodone/Acetaminophen 5mg/325mg, Hydromorphone 2mg, or Tramadol 50mg) every 4 hours and 800 mg Motrin for 10 days every 8 hours as needed for moderate to severe pain (4-10 on numeric rating scale).
  Interventions: Drug: Motrin and narcotic

INTERVENTIONS:
Drug: Motrin and narcotic — See described earlier

SUMMARY:
The aim of this study is to determine feasibility of a randomized controlled trial and estimates of efficacy for pain control of a scheduled pain regimen versus an as needed pain regimen for participants undergoing same day surgery procedures.

ELIGIBILITY:
Inclusion Criteria:

* Any outpatient surgeries performed at Cape Fear Valley Medical Center by Dr. Van Fossen during the duration of the study, including: laparoscopic cholecystectomy, laparoscopic appendectomy, laparoscopic ventral/umbilical/incisional hernia repair, open ventral/umbilical/incisional hernia repair, laparoscopic inguinal hernia repair, open inguinal hernia repair, lumpectomy, sentinel lymph node biopsy, lymph node biopsy, mass excision skin or subcutaneous, diagnostic laparoscopy, laparoscopic lysis of adhesions, pilonidal cyst excision, hemorrhoidectomy, anal fissure/sphincterotomy, anal fistulectomy, rectal exam under anesthesia, wound debridement, and wound closure
* Outpatients who are medically eligible to receive the standard post surgery medication protocol (the scheduled pain protocol used in this study).
* Age 18-65

Exclusion Criteria:

* Participants with the following conditions will be excluded from our study: fibromyalgia, chronic pain, cancer (except for breast cancer). This is because these participants have pain at baseline and it will be difficult to discern if their pain is from surgery or their chronic condition.
* Participants on chronic pain medications will also be excluded from our study because it will be difficult to tell if their pain control is related to their established regimen or the one we are implementing.
* If participants who are not fluent in English, because all study materials are in English.
* Participants with stage 3 Chronic Kidney Disease or higher will also be excluded from the study as they cannot take ibuprofen (according to National Kidney Foundation), which is included in our pain regimen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of trial | 2 weeks
  To measure feasibility of the study, the following data will be collected:
  1. Number of participants eligible for the study
  2. Number of participants contacted about the study
  3. Number of participants consented
  4. Number of participants being at least 80% adherent to medication protocol
  5. Number of drop-outs in the study and reason for drop out
  6. Number of Adverse Events reported to study personnel. For all non-consented participants, only counts will be included (e.g., 5 participants who refused to consent), no identifying or private information will be collected.

SECONDARY OUTCOMES:
Estimate of effect size pain control | 2 weeks
  Daily diary of pain (10 point scale)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Van Fossen, DO, Principal Investigator — Cape Fear Valley Health
Locations (1):
- Cape Fear Valley Medical Center, Fayetteville, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No